CLINICAL TRIAL: NCT06857565
Title: Interventional Study on Efficacy of Lactobacillus Crispatus M247 in Prevention and Treatment of Recurrent URinary Tract Infections in Association With Supplementation With Enterococcus Faecium L3 and Bifidobacterium Animalis Subsp. Lactis BB-12 (URTI): A Controlled Randomized Pilot Clinical Trial
Brief Title: Study to Evaluate the Efficacy of Lactobacillus Crispatus M247 in the Prevention and Treatment of Recurrent Urinary Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental medicine, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0038288/22/07.12.2022
Record Dates: First submitted 2025-02-22; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Recurrent Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, open-label study assessing the efficacy of Lactobacillus crispatus M247 (CRISPACT®) in preventing recurrent urinary tract infections (rUTIs) in women with a history of recurrent UTIs. Participants will be assigned to either the Probiotic Group, receiving CRISPACT® plus iNatal-duo®, or the Control Group, receiving iNatal-duo® alone. The primary outcome is the reduction in UTI recurrence over 12 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRISPACT® Group (Experimental): Participants in this group will receive iNatal-duo® (containing Bifidobacterium animalis subsp. lactis BB-12 and Enterococcus faecium L3) 1 sachet per day orally for 30 days, along with CRISPACT® (Lactobacillus crispatus M247) administered both orally and vaginally for 90 days. The intervention aims to assess whether probiotic therapy reduces the frequency and severity of recurrent urinary tract infections (rUTIs) over 12 months compared to standard treatment.
  Interventions: Dietary Supplement: Lactobacillus crispatus M247; Dietary Supplement: iNatal-duo® (containing Bifidobacterium animalis subsp. lactis BB-12 and Enterococcus faecium L3)
- Control Group (Active Comparator): Participants in this group will receive iNatal-duo® alone 1 sachet per day orally for 30 days without additional probiotic supplementation. This group will serve as a control to evaluate the comparative effectiveness of probiotic supplementation in preventing rUTI recurrence.
  Interventions: Dietary Supplement: iNatal-duo® (containing Bifidobacterium animalis subsp. lactis BB-12 and Enterococcus faecium L3)

INTERVENTIONS:
Dietary Supplement: Lactobacillus crispatus M247 — CRISPACT® (Lactobacillus crispatus M247), Pharmextracta, S.p.A
  Arms: CRISPACT® Group
Dietary Supplement: iNatal-duo® (containing Bifidobacterium animalis subsp. lactis BB-12 and Enterococcus faecium L3) — iNatal-duo®, PharmExtracta S.p.A

SUMMARY:
This randomized, open-label, controlled clinical trial evaluates the efficacy and safety of Lactobacillus crispatus M247 (CRISPACT®) in preventing recurrent urinary tract infections (rUTIs) in women. The study will enroll 130 adult female participants with a history of recurrent UTIs, defined as ≥3 episodes in the past year or ≥2 episodes in the past six months. Participants will be randomized into two groups: the Probiotic Group, receiving iNatal-duo® (containing Bifidobacterium animalis subsp. lactis BB-12 and Enterococcus faecium L3) for 30 days, plus CRISPACT® (Lactobacillus crispatus M247) for 90 days; and the Control Group, receiving iNatal-duo® alone for 30 days without additional probiotic supplementation. The primary outcome is a reduction in the frequency and severity of rUTIs over 12 months, while secondary outcomes include symptom improvement, impact on quality of life, and safety assessments.

DETAILED DESCRIPTION:
Recurrent urinary tract infections (rUTIs) represent a significant public health issue, disproportionately affecting women with hormonal fluctuations, sexual activity-related risks, or previous antibiotic use. Standard treatment involves antibiotic therapy, which, while effective, contributes to antimicrobial resistance, gut microbiota imbalances, and increased recurrence risk. Probiotics, particularly Lactobacillus crispatus, have been shown to restore vaginal microbiota balance, prevent uropathogen overgrowth, and reduce the likelihood of rUTIs. This study aims to assess whether CRISPACT® (Lactobacillus crispatus M247), administered orally and vaginally, provides superior protection against rUTIs compared to standard care with iNatal-duo® alone.

The study will follow a randomized, controlled design with 130 participants divided into two arms. The Probiotic Group will receive iNatal-duo® for 30 days, combined with CRISPACT® (Lactobacillus crispatus M247) for 90 days, while the Control Group will receive iNatal-duo® alone for 30 days without additional probiotic supplementation. The primary objective is to evaluate the reduction in UTI recurrence over 12 months, measured through clinical diagnoses and patient-reported data. Secondary objectives include evaluating symptom relief, patient-reported quality of life improvements (EQ-5D, King's Health Questionnaire), and the safety and tolerability of probiotic therapy. The study seeks to provide scientific evidence for integrating probiotics into rUTI prevention strategies, reducing antibiotic dependence, and improving women's urogenital health.

ELIGIBILITY:
Inclusion Criteria:

* History of recurrent urinary tract infections (rUTIs) with at least 3 episodes per year.
* No antibiotic treatment in the past 4 weeks before enrollment.
* Not currently pregnant or breastfeeding.
* Willing to provide vaginal and urine samples for microbiota analysis.
* Able to provide informed consent and comply with study procedures.

Exclusion Criteria:

* Current urinary tract infection (UTI) at the time of enrollment.
* Use of immunosuppressive therapy or presence of immunodeficiency disorders.
* Use of other probiotics within 4 weeks before enrollment.
* Known allergy or hypersensitivity to study products (Lactobacillus crispatus M247 or iNatal-duo®).
* History of pelvic radiation therapy or major gynecological surgery.
* Severe gastrointestinal conditions, including inflammatory bowel disease.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since the study focuses on recurrent urinary tract infections, which are more prevalent in women.
Enrollment: 130 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Recurrent Urinary Tract Infections (rUTIs) | 12 months
  The primary outcome will assess the recurrence rate of urinary tract infections over 12 months in participants receiving CRISPACT® (Lactobacillus crispatus M247) + iNatal-duo® compared to those receiving iNatal-duo® alone. A lower recurrence rate in the intervention group will indicate efficacy in preventing rUTIs.

SECONDARY OUTCOMES:
Change in Vaginal Microbiota Composition | Baseline, 3 months, 12 months
  This outcome will evaluate shifts in vaginal microbiota composition, particularly the prevalence of Lactobacillus crispatus, before and after intervention.
Change in Antibiotic Use for UTIs | 12 months
  The number of antibiotic courses required to manage rUTIs will be recorded, comparing the probiotic intervention group to the control group.
Change in urinary discomfort | Baseline, 6 months, 12 months
  Assessment tool: Visual Analog Scale (VAS) Scale: 0 = No discomfort, 10 = Worst imaginable discomfort
Change in pain severity | Baseline, 6 months, 12 months
  Assessment tool: Visual Analog Scale (VAS) Scale: 0 = No pain, 10 = Worst imaginable pain
Change in overall well-being | Baseline, 6 months, 12 months
  Assessment tool: SF-36 Quality of Life Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Medicine & Technological Innovation Dept. University of Insubria, Varese, Italy

IPD SHARING:
Plan to Share IPD: No